CLINICAL TRIAL: NCT03522168
Title: Pediatric Trials Network Long-term Antipsychotic Pediatric Safety Trial (LAPS) NICHD-2016-LAP01 Phase 4 Trial
Brief Title: Long-term Antipsychotic Pediatric Safety Trial
Acronym: LAPS
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Daniel Benjamin, Kiser-Arena Professor of Pediatrics, Duke University
Other Study IDs: Pro00084468
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Weight, Body
MeSH Terms: conditions — Body Weight | interventions — Risperidone; Aripiprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Main Trial: Obtain whole blood samples for future genetic analyses that may be used to determine if there are any genetic factors that might be used to personalize risk assessments.
  Registry Sub-Study: None.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Risperidone group: Risperidone, n=350, including 30 children 3 - <6 years old and 320 children 6 - <18 years old. ~50% - ~80% of the entire group will have <90 days of prior treatment with any antipsychotic.
  Interventions: Drug: Risperidone
- Aripiprazole group: Aripiprazole group, n=350, including 30 children 3 - <6 years old and 320 children 6 - <18 years old. ~50% - ~80% of the entire group will have ≤90 days of prior treatment with any antipsychotic.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Risperidone — Medications prescribed as standard of care for Schizophrenia, Bipolar mania/acute treatment of manic and mixed episodes associated with Bipolar I disorder, Tourette's disorder, persistent (chronic) motor or vocal tic disorder and Irritability associated with autistic disorder
  Other Names: Risperdal
  Groups: Risperidone group
Drug: Aripiprazole — Medications prescribed as standard of care for Schizophrenia, Bipolar mania/acute treatment of manic and mixed episodes associated with Bipolar I disorder, Tourette's disorder, persistent (chronic) motor or vocal tic disorder and Irritability associated with autistic disorder
  Other Names: Abilify
  Groups: Aripiprazole group

SUMMARY:
Main LAP01 study: The purpose is to evaluate the long-term pathologic weight changes associated with multi-year risperidone or aripiprazole therapy in 3 - <18-year-old children, who have varying durations of prior antipsychotic drug exposure from the start of study Month 0 (M0). This is critical because children appear to have greater vulnerability to antipsychotic-associated weight gain than adults, and obesity has significant effects on morbidity and mortality.

An additional sub-study (registry sub-study) was added via a protocol amendment. This registry sub-study is optional for participants and only participants who participate in the main study are eligible if they were 6 to less than 18 years of age at the time of the M0 visit. Participants who consent to this registry sub-study will participate in yearly in-person visits and complete monthly assessments remotely over the course of two additional years from the time of their final visit of the main LAP01 study.

DETAILED DESCRIPTION:
Main LAP01 study: Prospective, multi-site, Phase 4, longitudinal observational study designed to systematically collect robust longitudinal post-marketing safety and quality of life data about multi-year pediatric treatment with risperidone or aripiprazole. Screening may occur for up to 37 days prior to enrollment. Assessments will occur at in-person visits planned at months 0, 6, 12, 18 and 24, and at unscheduled, in-person visits that study staff request when the participant switches or stops antipsychotic monotherapy with risperidone or aripiprazole, adds or stops treatment with a weight modifying agent, becomes pregnant, chooses to withdraw from the study prematurely or, has an ongoing Serious Adverse Event (SAE) that requires further assessment. Monthly remote interim contacts occurring between in-person visits will monitor for changes (other than dose related) in antipsychotic therapy or weight modifying treatments, potential SAEs, and potential pregnancy. The participant, his/her parent/guardian, and the participant's personal psychotropic-prescribing medical provider (PPPMP) will make any and all decisions related to antipsychotic medications, any other medications, and the participant's current mental state, developmental/psychiatric condition, and level of risk for potential harm to self or others independent of the study procedures and assessments. Study staff (SS) will share with the participant's PPPMP all lab results and changes in the participant's AEs or clinical presentation, which the study medical clinician (SMC) considers medically concerning based on the participant's assessment during in-person visits. If an emergency safety concern is evident during an in-person visit, the SMC will immediately assess the participant, following medical standard-of-care procedures, to determine whether the participant is safe to leave the clinic or requires additional emergency care. If new or worsening symptoms are reported by the participant or parent/guardian during remote interim contacts, the participant and/or parent/guardian will be instructed to contact the PPPMP directly.

Registry sub-study: Participants who choose to participate will consent via a mobile application (Pattern Health) and will measure their height and weight at home monthly (also collected through the Pattern Health mobile application). One questionnaire will be completed every 6 months via the Pattern Health mobile application. Yearly in-person visits will be conducted to obtain in-clinic height, weight, vital signs and review concomitant medications.

ELIGIBILITY:
Main Study

Inclusion Criteria:

1. Parent/guardian has provided informed consent
2. Participant has provided assent if developmentally appropriate and as required by the institutional review board (IRB)
3. 3 - <18 years of age inclusive at time of M0 visit
4. Participant, when developmentally appropriate, and parent/guardian are:

   1. Willing to authorize exchange of information between the SS and the participant's PPPMP and/or other significant medical provider
   2. Affirm participant's use at M0 visit of either risperidone or aripiprazole mono-antipsychotic therapy as prescribed by participant's PPPMP
5. Based on their age at the time of M0 visit, participant is receiving aripiprazole or risperidone at the dose and for the diagnoses as listed below:

   1. Participants ages 3 - < 6 years can have any diagnosis and any dose
   2. Participants ages ≥ 6 - <18 years at the doses and for the diagnoses listed below

      Labeled Indications (Closely Related Disorders)

      Aripiprazole 2-30 mg/day
      * Irritability associated with autistic disorder:

      (Irritability in autism spectrum disorder) - Treatment of Tourette's disorder: (Tourette's disorder, persistent (chronic) motor or vocal tic disorder)

      - Bipolar mania/acute treatment of manic and mixed episodes associated with Bipolar l disorder: (Bipolar spectrum disorders including disruptive mood dysregulation disorder)

      - Schizophrenia: (Schizophrenia spectrum disorders including schizoaffective disorder, psychosis not otherwise specified, and delusional disorder)

      Risperidone 0.25-6 mg/day - Irritability associated with autistic disorder: (Irritability in autism spectrum disorder)

      - Bipolar Mania: (Bipolar spectrum disorders including disruptive mood dysregulation disorder)

      - Schizophrenia: (Schizophrenia spectrum disorders including schizoaffective disorder, psychosis not otherwise specified, and delusional disorder)
      * MYCITE® (aripiprazole) and all forms of injectables are not permitted in this study
6. Guardian anticipates risperidone or aripiprazole treatment will continue for ≥6 months

Exclusion Criteria:

1. History of prior or current diagnosis of an eating disorder or meets diagnostic criteria for an eating disorder as described in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and determined by psychiatric exam
2. Pre-existing or suspected major medical, metabolic, or genetic condition that is expected to be associated with weight, cardiovascular, neuromotor, or endocrine problems
3. Known or self-reported pregnancy
4. Taking antipsychotic medication other than either risperidone or aripiprazole at the time of M0 visit
5. Contraindications to participation in the study in the opinion of the SMC
6. Unwilling or unable to provide back-up family contact information

Registry Sub-Study

Inclusion Criteria:

1. Enrolled in LAPS Trial
2. Access to a personal mobile device (with Bluetooth capability and data or internet access) and willing to use it for the purposes of this study
3. Parent/guardian/LAR/participant has provided informed consent
4. Participant has provided assent/consent if developmentally appropriate and as required by the institutional review board (IRB)
5. Participant was part of the 6 to <18 year-old group in the LAPS Trial

Exclusion Criteria:

1. Participant has completed the M24 LAPS Trial Visit

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Main Study:
  The study population will consist of two groups of children 3 - <18 yrs old at the M0 visit:
  * Risperidone group, n=350, including 30 children 3 - <6 yrs old and 320 children 6 - <18 yrs old, ~ 50% - 80% will have <90 days of prior treatment with any antipsychotic.
  * Aripiprazole group, n=350, including 30 children 3 - <6 yrs old and 320 children 6 - <18 yrs old., ~ 50% - 80% will have ≤90 days of prior treatment with any antipsychotic.
  We will target participants within each treatment group to be distributed across the age range to permit analyses of age effects with:
  * ~30 being 3 - <6 years
  * ≥35% (n ≥123) being 6 - <12 years
  * ≥35% (n ≥123) being 12 - <18 years PK sub group at selected sites includes 24 participates, details in protocol.
  Registry Sub-Study Registry participants will be selected exclusively from the population that has enrolled onto the LAPS Trial.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Main Trial: Change in BMI z-score | Baseline, 24 months
  Longitudinally, evaluate the long term pathologic weight changes associated with multi- year risperidone or aripiprazole therapy over a period of 24 months in children ages 3 -<18 years with varying durations of prior antipsychotic drug exposure at the M0 visit. The primary analysis will focus on changes in the modified Body Mass Index (BMI) z- score in children 6 - <18 years old from M0 visit over 24 months of follow up.
Registry Sub-Study: Modified Body Mass Index (BMI) z-score | Up to 24 months
  Evaluate the long-term pathologic weight changes associated with multi-year risperidone or aripiprazole therapy over a period of 24 to 50 months in children who were 6 to <18 years of age at the time of LAPS Trial enrollment

SECONDARY OUTCOMES:
Main Trial: Measure of weight change | Baseline, 24 months
  Change in BMI category and Modified BMI z-score increase of ≥1.0 unit from M0
Main Trial: Metabolic measures associated with risk of diabetes and cardiovascular disease | Baseline, 24 months
  Clinical laboratory evaluations for high-sensitivity C-reactive protein (hs-CRP); hemoglobin A1c (Hgb A1c); Presence of acanthosis nigricans or, in females only, hirsuitism on physical exam
Main Trial: Prolactin related outcomes | Baseline, 24 months
  Clinical laboratory evaluation of serum prolactin; Incidence of gynecomastia in males on physical exam
Main Trial: Uniformly Elicited Events of Special Interest | Baseline, 24 months
  A standardized semi-structured interview will be used by the SMC to assess events of special interest in all participants at every in-person visit [56]. The form queries for potential hospitalizations, emergency department visits, and urgent care visits and for pregnancy. The form also evaluates frequent or especially concerning adverse effects seen with antipsychotics including behavioral events. Targeted symptoms are: Sedation, Increased sleep, Problems with attention, thinking or learning Insomnia, Arrhythmias, Light-headedness (Orthostasis vs Vertigo), Seizures, Increased appetite, Decreased appetite, Tics, Tremors, Parkinsonian symptoms, Akathisia, Drooling, Dyskinesia, Polydipsia, Polyuria, Enuresis, Galactorrhea, Amenorrhea, Sexual dysfunction/anorgasmia, Diabetes, Fractures Menorrhagia, Lack of satiety
Main Trial: Adverse effects | Baseline, 24 months
  Serious adverse events Adverse events (AEs) of mild (grade 1) severity and related to risperidone or aripiprazole All adverse events of moderate (grade 2) severity or greater regardless of relatedness to risperidone or aripiprazole
Main Trial: Suicidality | Baseline, 24 months
  Assessed using DASS
Main Trial: Neuromotor effects | Baseline, 24 months
  Abnormal Involuntary Movement Scale (AIMS) Simpson Angus Extrapyramidal Symptoms Scale (SAS)
Main Trial: AEs (Adverse Events) | Baseline, 24 months
  Elicited AEs, including AEs of mild (grade 1) and related to risperidone or aripiprazole, and all AEs of moderate (grade 2) or greater and clinically significant changes in suicidality.
Main Trial: Pediatric Quality of Life Inventory | Baseline, 24 months
  Relationship of risperidone or aripiprazole therapy to adaptive functioning and quality of life as assessed by the Pediatric Quality of Life Inventory (PedsQL, 23 item), and changes in the intensity or frequency of pre-existing behavioral problems indicated at M0 (baseline). The 23-item PedsQL Generic Core Scales were designed to measure the core dimensions of health as delineated by the World Health Organization in individuals aged 2 years and older. The main scales include physical functioning, emotional functioning, social functioning, and school functioning. Summary scores can also be utilized to measure change over time on a five point scale for 0 = "Never a Problem" to 5 = "Almost Always a Problem". The guardian will be asked to complete the parent version for reporting on their child's quality of life.
Main Trial: School and Work Questionnaire (SWQ) | Baseline, 24 months
  Relationship of risperidone or aripiprazole therapy with age-appropriate skip patterns, school promotions and graduations, changes in school supports, type of living situations, romantic relationships, arrests, and types and extent of employment during the interval since the prior assessment.
Main Trial: Caregiver Strain Questionnaire (CSQ) | Baseline, 24 months
  Relationship of risperidone or aripiprazole therapy to adaptive functioning and quality of life as assessed ) by the Caregiver Strain Questionnaire (CSQ) and changes in the intensity or frequency of pre-existing behavioral problems indicated at M0 (baseline). This is a 21-item questionnaire with a categorical scale ranging from 1 (not at all a problem) to 5 (very much a problem) that assesses the caregiver's quality of life. It asks specifically about the caregiver's quality of life by assessing the impact of caring for a child with emotional and behavioral problems. The questions include information about disruption of family life and relationships; demands on time; negative, mental, and physical health effects for any family member; financial strain; feelings of sacrifice; disruption of social/community life; worry/guilt; fatigue/strain; and embarrassment.
Main Trial: Delighted-Terrible Faces Scale (DTFS) | Baseline, 24 months
  Relationship of risperidone or aripiprazole therapy to adaptive functioning and quality of life as assessed by the Delighted-Terrible Faces Scale (DTFS) and changes in the intensity or frequency of pre-existing behavioral problems indicated at M0 (baseline). The DTFS is a uni-dimensional, single item scale that will be used to assess the participant's perceived life quality. Faces expressing various feelings are depicted, and the participant is asked which face comes closest to expressing how he/she feels about his/her life over the past month. The participant can then select from the range of seven categorical faces depicting from one-delighted to seven-terrible expressions. This scale is included because it can be easily completed by participants with limited verbal and cognitive abilities as well as by very young children.
Main Trial: PK CL/F | 24 months
  CL/F, apparent total clearance of the drug from plasma after oral administration at steady state
Main Trial: PK Vss/F | 24 months
  Vss/F, apparent volume of distribution at steady state after non-intravenous administration at steady state
Main Trial: PK AUCss | 24 months
  AUCss, area under the curve at steady state
Main Trial: PK Cmax | 24 months
  Cmax, maximum concentration at steady state
Main Trial: PK Tmax | 24 months
  Tmax, time of maximum concentration at steady state
Main Trial: PK T1/2 | 24 months
  T1/2, half-life at steady state
Registry Sub-Study: Parent/guardian/former guardian/LAR completed Pediatric Quality of Life Inventory (PedsQL, 23 item) survey. | Up to 24 months
  Change in PedsQL outcomes over time from M0 LAPS Trial in-person visit to R24 LAPS Registry mobile data collection

OTHER OUTCOMES:
Registry Sub-Study: Weight and height | Up to 24 months
  Concordance between weight and height collected over time from R0 LAPS Registry to R24 LAPS Registry in-person visits and mobile data
Registry Sub-Study: Demographics, Measurements and Vital Signs, Lab Measurements, Clinical data | Up to 24 months
  * Describe extraction and transfer completeness of proposed data elements (e.g. blank fields versus error fields).
  * Describe if extracted measurements, vital signs, and lab values are within the expected biological range.
  * Describe concordance of extracted height and weight values with height and weight values obtained from in-person study visits.
  * Describe the format and usability of extracted data.

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — Duke Clinical Research Institution (DCRI); Kevin Watt, MD, PhD, Principal Investigator — University of Utah; Karan Kumar, MD, MS, Principal Investigator — Duke Clinical Research Institution (DCRI)
Locations (37):
- United States (37):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - OM Research, Lancaster, California
  - UCLA Semel Institute, Los Angeles, California
  - Yale Child Study Center, New Haven, Connecticut
  - Clinical Trials Solution, Miami, Florida
  - South Florida Behavioral Health Network, Miami, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Valley Healthcare System, Columbus, Georgia
  - IACT Health, Grayson, Georgia
  - Attalla Consultants LLC dba Institute for Behavioral Medicine, Smyrna, Georgia
  - AMR-Baber Research, Inc., Naperville, Illinois
  - Beacon Medical Group, South Bend, Indiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Lurie Center for Autism, Lexington, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield, Michigan
  - Pine Rest Christian Mental Health Services, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Child and Family Study Center, Durham, North Carolina
  - Behavioral Health Hospital Oupatient Clinic, Greensboro, North Carolina
  - Cone Health Outpatient Behavioral Health, Greensboro, North Carolina
  - Carolina Partners in Mental HealthCare, PLLC, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Avera McKennan University Psychiatry Associates, Sioux Falls, South Dakota
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - BioBehavioral Research of Austin, Austin, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Neuropsychiatric Associates, Woodstock, Vermont
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All data collected is uploaded into the National Institute of Health data repository (DASH) at the end of the study (de-identified).
Time Frame: Data will be uploaded to the repository within 2 years of study completion. It will be maintained in the repository indefinitely.
Access Criteria: In order to have access, researchers have to complete a Data access request. NICHD will review the request and either approve or deny it. IRB approval must be obtained by the researcher to access the data.
  https://dash.nichd.nih.gov/Resource/DataRequestChecklist
URL: https://dash.nichd.nih.gov/

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT03522168/Prot_001.pdf
  • Informed Consent Form (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT03522168/ICF_002.pdf